CLINICAL TRIAL: NCT04134273
Title: A Randomized, Double-Blind, Multiple Center Placebo Controlled Study Comparing Taro Product to RLD and Both Treatments to a Placebo Control in the Treatment of Acne Vulgaris.
Brief Title: Bio-equivalence Study With Clinical Endpoints in the Treatment of Acne Vulgaris
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sun Pharmaceutical Industries, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLPG 1809
Record Dates: First submitted 2019-10-18; First posted 2019-10-22 (Actual); Last update posted 2019-10-22 (Actual); Status verified 2019-10

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — Clindamycin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- CLPG Topical Gel 1% (Experimental): Clindamycin Phosphate Topical Gel 1%, applied to the face twice a day for 84 days.
  Interventions: Drug: CLPG Topical Gel 1%
- Clindamycin Phosphate Topical Gel 1% (Active Comparator): Clindamycin Phosphate Topical Gel 1%, applied to the face twice a day for 84 days.
  Interventions: Drug: Clindamycin
- Vehicle of the test product (Placebo Comparator): Placebo (vehicle of the test product), applied to the face twice a day for 84 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CLPG Topical Gel 1% — Clindamycin Phosphate Topical Gel 1% (Taro Pharmaceuticals U.S.A, Inc.)
  Other Names: Topical Gel 1%
  Arms: CLPG Topical Gel 1%
Drug: Clindamycin — Clindamycin Phosphate topical gel 1%
  Other Names: Topical Gel 1%
  Arms: Clindamycin Phosphate Topical Gel 1%
Drug: Placebo — Placebo (vehicle of the test product) (Taro Pharmaceuticals Inc.)
  Other Names: Vehicle
  Arms: Vehicle of the test product

SUMMARY:
This study is to evaluate the therapeutic equivalence and safety of Taro Product to RLD in the treatment of acne vulgaris.

DETAILED DESCRIPTION:
The study objectives are to evaluate the therapeutic equivalence and safety of Taro Product to RLD in the treatment of acne vulgaris and to demonstrate the superiority of the efficacy of the test and reference products over the placebo control.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or non-pregnant female aged ≥ 12 and ≤ 40 years with a clinical diagnosis of acne vulgaris
* Subjects who are 18 years of age or older (up to the age of 40) must have provided IRB approved written informed consent. Subjects 12 to 17 years of age, inclusive, must have provided IRB approved written assent; this written assent must be accompanied by an IRB approved written informed consent from the Subject's legally acceptable representative (i.e., parent or guardian).
* Subjects must have a definite clinical diagnosis of acne vulgaris severity grade 2, 3, or 4 as per the Investigator's Global Assessment (IGA).

Exclusion Criteria:

* Female Subjects who are pregnant, nursing or planning to become pregnant during study participation.
* Subjects with a known hypersensitivity to clindamycin or lincomycin and/or any ingredients in the study drugs.
* Subjects with the presence of any skin condition that would interfere with the diagnosis or assessment of acne vulgaris (e.g., on the face: rosacea, dermatitis, psoriasis, squamous cell carcinoma, eczema, acneiform eruptions caused by medications, steroid acne, steroid folliculitis, or bacterial folliculitis).

Ages: 12 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1260 (Actual)
Dates: Start 2019-03-20 (Actual); Primary Completion 2019-09-17 (Actual); Study Completion 2019-10-15 (Actual)

PRIMARY OUTCOMES:
Demonstration of Bioequivalence | Week 12
  Demonstration of Bioequivalence in percent change in inflammatory and non-inflammatory lesion counts.

CONTACTS AND LOCATIONS:
Locations (1):
- Catawba Research, LLC, Charlotte, North Carolina, United States